CLINICAL TRIAL: NCT06454864
Title: Multiple Risk Factor Intervention Trial In Breast Cancer Survivors
Acronym: MsFITBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB #45301
Record Dates: First submitted 2024-05-22; First posted 2024-06-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Disturbance; Sedentary Behavior; Breast Cancer Female
MeSH Terms: conditions — Sedentary Behavior | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: 3-arm parallel-group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind participants to their assigned intervention. Care providers are not involved. The outcome assessors for any assessments involving potential for subjectivity in data collection or analysis will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guidelines-based physical activity (Experimental): 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening.
  Interventions: Behavioral: Guidelines-based physical activity
- Guidelines-based physical activity and healthy eating (Experimental): Arm Description: 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening + counselling to follow Canada's Food Guide.
  Interventions: Behavioral: Guidelines-based healthy eating; Behavioral: Guidelines-based physical activity
- Stretching exercise (Placebo Comparator): Whole-body stretching.
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Guidelines-based healthy eating — One-on-one phone/virtual counselling from a registered dietitian to change dietary habits to be in line with Canada's Food Guide.
  Arms: Guidelines-based physical activity and healthy eating
Behavioral: Guidelines-based physical activity — Through a combination of exercise trainer-led in-person and virtual sessions, as well as counselling for independent aerobic exercise, participants will be guided to achieve 150 weekly minutes of moderate-intensity aerobic activity and twice weekly whole-body muscle strengthening.
  Arms: Guidelines-based physical activity; Guidelines-based physical activity and healthy eating
Behavioral: Stretching exercise — Twice weekly virtual instructor-led whole-body stretching.
  Arms: Stretching exercise

SUMMARY:
This study aims to produce new evidence on the efficacy of exercise and diet for cardiometabolic risk reduction in BC survivors. Using a 3-arm RCT with to 6 months of 1) exercise following Health Canada guidelines; 2) the same exercise plus counselling to follow Canada's Dietary Guidelines to improve diet quality; or 3) stretching group, this study will answer the following questions:

* What is the impact of exercise on cardiometabolic health and body composition in BC survivors?
* What is the effect modification of adding a diet quality intervention to exercise on cardiometabolic health and body composition?
* Is there a link between the capacity of skeletal muscle adaptation to exercise (and diet) and insulin resistance in BC survivors?

The investigators hypothesize that: 1) exercise will improve cardiometabolic and body composition outcomes 2) improvements in cardiometabolic outcomes will be enhanced by the addition of diet quality, which will be essential or additive for Matsuda index, metabolic syndrome, Framingham CVD risk, thigh myosteatosis, muscle mass, VO2peak, 3) skeletal muscle insulin signalling transduction will be impaired in BC survivors via dampened expression of insulin-responsive proteins (e.g. GLUT4) and co-occur with impaired muscle quality (e.g., higher rates of fat depots, presence of fibrous tissue) negatively impacting insulin signalling.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Diagnosis of stage I, II, or III breast cancer, post-menopausal at the time of diagnosis (haven't had a menstrual cycle within 12 months or greater)
* Receipt of aromatase inhibitors for 12 months or more in the past, but do not have to be currently on aromatase inhibitors.
* Willing and able to complete all study assessments
* BMI ≥ 25 kg/m2
* Able to commit to come to the University once per week for 24 weeks.

Exclusion Criteria:

* Received chemotherapy within the past 11 months
* Diagnosed with metastatic cancer
* Currently taking tamoxifen
* Currently receiving chemotherapy, targeted therapy or radiation treatment
* Distant recurrence or diagnosis of metastatic cancer since early-stage breast cancer diagnosis
* Diagnosed cardiovascular diseases, type 2 diabetes, non-alcoholic fatty liver disease, uncontrolled thyroid condition, or respiratory disease (e.g., COPD or severe or uncontrolled asthma).
* Major signs or symptoms of cardiovascular diseases, diabetes, or renal disease (taken from the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription 11th edition Table 2.1: pain or discomfort in the chest, neck, jaw, arms with rest or exercise, shortness of breath at rest or with mild exertion, dizziness or syncope, loss of balance or passing out, ankle edema, palpitations or tachycardia, intermittent claudication, known heart murmur, unusual fatigue with usual activities.)
* American Heart Association's absolute or relative contraindications for symptom-limited maximal exercise testing (myocardial infarction, aortic or coronary artery stenosis, heart failure, pulmonary embolism or deep vein thrombosis, inflammation of the heart (myocarditis, pericarditis, and/or endocarditis), uncontrolled cardiac arrhythmia, advanced or complete electrical heart block, stroke or transient ischemia attack, blood pressure >200mmHg/100mmHg, a cancer diagnosis other than skin cancer)
* Unable to provide informed consent or communicate in English
* Pregnant or breast-feeding currently or in the past 3 months
* Mobility limitations to aerobic exercise (i.e., wheelchair, walker use, limp impeding walking)
* Smoking cigarettes or marijuana within the past 3 months
* Taking exogenous hormones in any format currently or in the past 3 months
* Contraindications to research MRI (e.g., pacemaker, magnetic implants)
* BMI exceeding 40 kg/m2
* Extreme claustrophobia
* Self-report >30 min/week of moderate-to-vigorous intensity aerobic physical activity
* Following a diet that largely restricts entire food groups or time of eating (e.g., vegan, ketogenic, carnivore, one meal a day) in last 3 months
* Experienced significant weight loss (i.e., >5 kg) in past 3 months
* Currently taking weight loss medications
* Diagnosed history of an eating disorder or self-report of potential undiagnosed eating disorder
* Plans to be away/unavailable for a substantial period of the intervention overall (i.e., >4 weeks throughout the 6 months or >2 weeks within the first 12 weeks of the intervention).
* Allergies to local anesthetics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 6 months
  As assessed by the Matsuda Index calculated from an oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Hepatic insulin resistance | 6 months
  Indirectly measured via HOMA-IR using fasting glucose and insulin levels
Metabolic syndrome severity | 6 months
  Calculated as a z-score to allow for tracking change in the interventions
Framingham 10-year risk (%) | 6 months
  Calculated using a widely-used standardized scoring system

OTHER OUTCOMES:
Cardiorespiratory fitness | 6 months
  Measured as peak volume of oxygen consumption via indirect calorimetry during a cardiopulmonary exercise test on a treadmill.
Heart Rate Recovery | 6 months
  Measured as the difference between peak heart rate during the cardiorespiratory fitness test and heart rate 2-minutes after stopping the exercise test.
avO2 difference | 6 months
  Calculated as the VO2 from the corresponding workload from the day 1 treadmill test divided by cardiac output at rest, submaximal, and maximal periods of the treadmill test
Blood Pressure | 6 months
  Measured as the average of the last 5 of 6 blood pressure measurements using an automatic blood pressure device.
Thigh Myosteatosis | 6 months
  Measured as thigh muscle fat fraction (percent of muscle compartment composed of fat pixels) determined from contiguous axial fat-water separation 3T magnetic resonance images of both thighs.
Knee flexion and extension (strength and endurance) | 6 months
  Measured using an isokinetic dynamometer (Biodex) to assess peak torque and total work in 30 repetitions of knee flexion.
Thigh Muscle Volume | 6 months
  Measured determined from contiguous axial fat-water separation 3T magnetic resonance images of both thighs
Concentration of biochemical markers of skeletal muscle protein content | 6 months
  Measured via western blotting from a skeletal muscle biopsy of the vastus lateralis muscle. Proteins of interest include those found in mitochondria, contractile signaling pathways, insulin signaling pathways, and in glucose and fat metabolism.
Concentration of biochemical markers of skeletal muscle structure | 6 months
  Measured via immunofluorescence from a skeletal muscle biopsy of the vastus lateralis muscle. Outcomes of interest will focus on indicators of histology of the skeletal muscle in withc a stain would include skeletal muscle capillarization, lipid content, and fiber type and cross-sectional area.
Concentration of biochemical markers of skeletal muscle enzyme activity | 6 months
  Measured via spectrophotometer to assess the maximal enzyme activity of enzymes involved in skeletal muscle oxidative capacity, from a biopsy of the vastus lateralis muscle.
Whole-body fat and fat-free mass | 6 months
  Measured using a body composition device (BodPod) to estimate whole body fat (in kg and %) and fat free mass (in kg and %).
Visceral adipose tissue | 6 months
  Volumes of adipose tissue in the visceral region measured using 3T fat-water separation magnetic resonance imaging
Liver fat fraction | 6 months
  Measured as percent of liver volume composed of fat pixels determined from 3 slices through the middle of the liver using the PROFIT1 3T magnetic resonance images sequence.
Body circumferences | 6 months
  Circumferences of the waist, hip and neck, measured using an inelastic tape
Lipid panel: HDL, LDL, total Cholesterol, Triglycerides | 6 months
  Analyzed from blood serum using a clinical assay at a core lab.
Hemoglobin A1c | 6 months
  Analyzed from blood plasma using a clinical assay at a core lab.
Dietary intake | 6 months
  Various components of dietary intake including macronutrients and micronutrients will be assessed through 3-day food records over 2 weekdays and 1 weekend collected using ASA-24 online system.
Liver enzymes: alanine transaminase (ALT), aspartate aminotransferase (AST), and albumin | 6 months
  Assessment of ALT, AST, and albumin via a fasting blood serum draw, analyzed on a clinical assay at a core lab.
Liver fibrosis | 6 months
  Liver T1 time evaluated using the PROFIT1 magnetic resonance sequence, validated marker of liver fibrosis.
Number of participants who met aerobic physical activity prescription | 6 months, 12 months
  Average adherence to prescribed aerobic physical activity weekly minutes measured via Garmin smartwatch
Number of participants who me the resistance exercise adherence | 6 months, 12 months
  Average adherence to prescribed resistance exercise activity weekly sessions via an attendance log
Diet quality | 3 months, 6 months, 12 months
  An overall measure of alignment with the dietary guidelines measured via the Healthy Eating Food Index-2019 calculated from 3-day diet records
Health-related quality of life | 3 months, 6 months, 12 months'
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100 and 2 component summary scales ranging from 0-50 with a higher score indicating better quality of life.
Breast Cancer specific related quality of life | 3 months, 6 months, 12 months'
  Assessed by EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
Psychosocial stress | 3 months, 6 months, 12 months'
  Assessed by the perceived stress scale (PSS-14) where individual scores can range from 0 to 56 with higher scores indicating higher perceived stress
Depression & Anxiety | 3 months, 6 months, 12 months'
  Measured by the Hospital Anxiety and Depression Scale (HADS); score ranges from 0-21 for each of depression and anxiety with a higher score indicating more severe depression or anxiety
Barriers and self-efficacy for physical activity | 3 months, 6 months, 12 months'
  Assessed by the barriers to self-efficacy scale (BARSE). For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100.
Physical activity motivation | 3 months, 6 months, 12 months'
  Assessed via the multi-process action control approach, which is a series of questionnaires developed to understand affective attitudes, instrumental attitudes, perceived capability over physical activity, perceived opportunity for physical activity, decisional intentions, behavioural regulation, physical activity habits, and identity around physical activity. Higher scores represent better physical activity motivations. (Reference: Rhodes, R.E. (2017). The evolving understanding of physical activity behavior: A multi-process action control approach. In A. J. Elliot (Ed), Advances in Motivation Science. (pp. 171-205).)
Sleep quality - subjective | 3 months, 6 months, 12 months'
  Subjectively assessed by the Pittsburgh Sleep Quality Index (PQSI), which measures components of sleep: sleep duration, disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use, with higher scores reflecting poorer sleep quality.
Sleep quantity and quality - device measured | 3 months, 6 months, 12 months'
  Measured via Garmin smartwatch for the total sleep duration and efficiency.
Self-reported physical activity | 3 months, 6 months, 12 months'
  Assessed by the Recent Physical Activity Questionnaire (RPAQ) that collects information about types and amounts of activity (sedentary and physical activities) over the last 3 months in the following domains: leisure time, occupation, commuting, domestic life, with greater scores indicating longer time engaging in forms of activity.
Hemoglobin | 6 months
  Assessed using a fasting blood plasma sample in a clinical assay at a core lab.
Concentration of free fatty acids | 6 months
  Assessed using fasting blood serum in a clinical assay.
Body weight | 6 months
  Assessed using a calibrated scale attached to the BodPod body composition device.
Body mass index (BMI) | 6 months
  Calculated from a measurement of height using a stadiometer and body weight (detailed above).
Energy Balance | 6 months
  Energy balance will be quantified as: 3-day avg calorie intake - [estimated resting metabolic rate + 3-day avg Garmin estimate of physical activity energy expenditure + 10% of calorie intake (thermic effect of food)].
Fatigue | baseline, 3 months, 6 months, 12 months'
  Assessed using the Multidimensional Fatigue Inventory (MFI-20), a 20-item self-assessment questionnaire that uses a 1 to 5 scale to indicate how statements regarding fatigue are representative of a respondent's experience. A higher score is indicative of higher levels of fatigue.
Risk of Type 2 Diabetes | baseline, 3 months, 6 months, 12 months'
  The online CANRISK tool (www.healthycanadians.gc.ca/en/canrisk) assigns scores to risk factors for type 2 diabetes (that overlap with cardiovascular disease/cancer), including age, body mass index, MVPA, fruit/vegetable intake, hypertension, pregnancy complications, ethnicity and education, and is validated for Canada's multiethnic population.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Kirkham, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No